CLINICAL TRIAL: NCT03114982
Title: Randomized, Double-blinded, Parallel-group, Exploratory Study to Assess The Immunogenicity and Safety of NBP608 and Varivax in Healthy Children
Brief Title: The Evaluation of Immunogenicity and Safety of NBP608 in Healthy Children 12 Months to 12 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP608_VZ_II_2015
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Varicella
Keywords: Prevention of varicella; Varicella-zoster vaccine
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low potency of NBP608 (Experimental): Single dose 0.5mL of low potency of NBP608 by subcutaneous injection into the outer aspect of the upper arm or the anterolateral thigh
  Interventions: Biological: NBP608
- Middle potency of NBP608 (Experimental): Single dose 0.5mL of middle potency of NBP608 by subcutaneous injection into the outer aspect of the upper arm or the anterolateral thigh
  Interventions: Biological: NBP608
- High potency of NBP608 (Experimental): Single dose 0.5mL of high potency of NBP608 by subcutaneous injection into the outer aspect of the upper arm or the anterolateral thigh
  Interventions: Biological: NBP608
- Varivax (Active Comparator): Single dose 0.5mL of Varivax by subcutaneous injection into the outer aspect of the upper arm or the anterolateral thigh
  Interventions: Biological: Varivax

INTERVENTIONS:
Biological: NBP608 — Preparation of the Oka/SK strain of live, attenuated varicella virus
  Arms: High potency of NBP608; Low potency of NBP608; Middle potency of NBP608
Biological: Varivax — Preparation of the Oka/Merck strain of live, attenuated varicella virus
  Arms: Varivax

SUMMARY:
This study evaluates the immunogenicity and safety of three different potencies of NBP608 and Varivax which are indicated for active immunization for the prevention of varicella. Total of 152 subjects (38 subjects per each treatment arm) of 12 months to 12 years of age are enrolled, and each subject is administered with single dose of vaccine which is randomly assigned.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blinded, active controlled, parallel-group study to evaluate the immunogenicity and safety of three different potencies of NBP608(low, middle, high potency) and Varivax which are indicated for active immunization for the prevention of varicella. Total of 152 subjects (38 subjects per each treatment arm) of 12 months to 12 years of age are enrolled, and each subject is administered with single dose of vaccine which is randomly assigned in 1:1:1:1 ratio. Stratified randomization for age group is used to achieve the balance of treatment assignment within age strata.

Total of four visits are scheduled including two visits via telephone contact. Blood sampling is conducted for immunogenicity assessment before and 6 weeks after vaccination at Visit 1 and Visit 3 respectively. Safety is monitored 1 week, 6 weeks and 26 weeks after vaccination through Visit 2*, Visit 3 and Visit 4* (*telephone contact)

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged between 12 months and 12 years old who are available for the follow-up during the study period
* After menarche females who are confirmed to be negative in a pregnancy test on the day of vaccination and agree to practice birth control for 3 months after the vaccination

Exclusion Criteria:

* Those with hypersensitivity to any component of the IPs(Investigational Products), such as gelatin or neomycin
* Those who have received a varicella vaccine previously
* Those with a history of hypersensitivity to vaccination, such as Guillain-Barre syndrome
* Those with congenital or acquired immunodeficiency
* Those with active untreated tuberculosis
* Those who have received or are expected to receive salicylates from 14 days prior to IP(Investigational Product) vaccination to Visit 3
* Those who have received or are expected to receive other vaccines from 1 month prior to IP(Investigational Product) to Visit 3
* Those who have received or are expected to receive other IPs(Investigational Products) in another clinical study from 1 month prior to IP(Investigational Product) vaccination to Visit 3

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate measured by FAMA(Fluorescent Antibody to Membrane Antigen) assay | 6 weeks after IP(Investigational Product) vaccination
  *FAMA(Fluorescent Antibody to Membrane Antigen) Seroconversion Rate: the rate of subjects who are converted from seronegative with FAMA(Fluorescent Antibody to Membrane Antigen) VZV(Varicella Zoster Virus) antibody titer < 1:4 before IP(Investigational Product) vaccination to seropositive with FAMA(Fluorescent Antibody to Membrane Antigen) VZV(Varicella Zoster Virus) antibody titer ≥ 1:4 at 6 weeks post-vaccination

SECONDARY OUTCOMES:
VZV (Varicella Zoster Virus) antibody GMT (Geometric Mean Titer) measured by FAMA(Fluorescent Antibody to Membrane Antigen) assay | 6 weeks after IP(Investigational Product) vaccination
VZV (Varicella Zoster Virus) antibody GMT (Geometric Mean Titer) measured by gpELISA (Glycoprotein Enzyme Linked Immunosorbent Assay) | 6 weeks after IP(Investigational Product) vaccination
Seroconversion rate measured by gpELISA (Glycoprotein Enzyme Linked Immunosorbent Assay) | 6 weeks after IP(Investigational Product) vaccination
  *gpELISA Seroconversion Rate : the rate of subjects who are converted from seronegative with < 50mIU/mL before IP vaccination to seropositive with ≥ 50mIU/mL at 6 weeks post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario Z. capeding, Dr, Principal Investigator — Research Institute for Tropical Medicine
Locations (1):
- Research Insitute for Torpical Medicine, Muntinlupa City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No